CLINICAL TRIAL: NCT06816121
Title: Identification and Validation of Blood-Based Biomarkers for Early Detection of Asymptomatic Lung Cancer in High-Risk Heavy Smokers
Status: Not yet recruiting | Type: Observational
Sponsor: Everest Detection, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RAD-01
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancers
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat samples derived from whole blood collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Non-Cancer Cohort: Patients With No Lung Nodules at Initial Computed Tomography (CT) Scan or Stable, Non-Suspicious Nodules at Follow-Up CT Scans
- Indeterminate Cohort: Patients with indeterminate pulmonary nodules actively in follow-up
- Highly Suspicious or Confirmed Lung Cancer Cohort: Patients with pathologic diagnosed, untreated lung cancer or highly suspicious for lung cancer that are still in workup
- "Other Cancer" Cohort: Patients with a pathologic diagnosis of cancers highly associated with smoking

SUMMARY:
The goal of this observational study is to develop and evaluate a blood test for asymptomatic heavy smokers to screen for those at highest risk of developing lung cancer. The aim of this study is to develop, train, and validate a blood-based screening test designed to detect biomarkers associated with lung cancer. The study will utilize samples collected from 4 distinct cohorts.

1. Participants confirmed to have lung cancer
2. Participants without cancer
3. Participants with moderate risk of lung cancer (indeterminate)
4. Participants confirmed to have other types of cancers linked to smoking

The main question this study aims to answer is whether the blood test can detect existing early-stage lung cancer in heavy smokers without symptoms and to provide insights into device performance and long-term outcomes when scans show no nodules, benign findings, or indeterminate nodules.

Participants will provide blood samples at the start of the study and during follow-up visits at 12 and 24 months. Participants will share information about their smoking history, lung cancer status, and relevant medical history

Researchers will collect blood samples, process them, and analyze the biomarkers at the Everest Detection laboratory. No results will be shared with participants or their doctors. The study will run for about 48 months, including a 24-month enrollment period and 24 months of follow-up to track participants' health and lung cancer outcomes.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Understands the study and can provide written informed consent
* Willing and able to provide a blood sample
* Age 30-80
* Current or former smoker

Non-Cancer Cohort:

* Recent CT scan within 3 months AND
* No lung nodules (Lung-RADS 1) or benign/stable nodules

Indeterminate Cohort:

* Recent CT scan within 12 months AND
* Indeterminate lung nodules under active monitoring

Highly Suspicious or Confirmed Lung Cancer Cohort:

* Confirmed untreated lung cancer OR
* Highly suspicious lung nodules undergoing diagnostic work-up

Other Cancer Cohort:

- Confirmed, untreated cancer associated with smoking

Exclusion Criteria:

* Cancer diagnosis within the last 5 years
* Systemic therapy, radiation, or surgery for cancer within 1 year prior to enrollment
* Any history of hematologic malignancies or myelodysplasia
* Known infection with HIV, HCV, or HBV
* Active pregnancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both smokers that meet USPSTF criteria for annual LD-CT screening (age 50-80, smoked >20 pack years, quit <15yr ago if former smoker) to younger (>30 years) and lighter smokers (>10 pack years)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker Discovery and Validation for Blood-Based Early Lung Cancer Detection in Heavy Smokers | From enrollment to the end of the study observation period of 24 months
  This study aims to discover and optimize biomarkers for a blood-based test that detects early-stage lung cancer in heavy smokers without symptoms. Researchers will develop and validate the test using blood samples from individuals with lung cancer, those at varying screening risk levels (Lung-RADS 1-4), and heavy smokers with smoking-related cancers.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to study-specific considerations and data use restrictions.